CLINICAL TRIAL: NCT00505063
Title: Phase II Prospective Trial of Vaccine Responses in Childhood Cancer Survivors
Brief Title: Prospective Trial of Vaccine Responses in Childhood Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-088
Record Dates: First submitted 2007-07-18; First posted 2007-07-20 (Estimated); Last update posted 2025-06-15 (Actual); Status verified 2024-06

CONDITIONS: Childhood Cancer; Multiple Diseases
Keywords: vaccine; childhood; cancer
MeSH Terms: conditions — Neoplasms | interventions — Vaccines; 13-valent pneumococcal vaccine; Measles-Mumps-Rubella Vaccine; Chickenpox Vaccine; Aging

ARMS (3):
- A (Other): Immunization Schedule patients <7 years.
  Interventions: Biological: Immunization Schedule patients <7 years.
- B (Other): Immunization Schedule patients > or = to 7 years and <11 years of age
  Interventions: Biological: Immunization Schedule patients > or = to 7 years and <11 years of age
- C (Other): Immunization Schedule patients > or = to 11 years of age
  Interventions: Biological: Immunization Schedule patients > or = to 11 years of age

INTERVENTIONS:
Biological: Immunization Schedule patients <7 years. — * Time 0 months: Prevnar 13 #1, Hib #1
  * Time 1 months: Pediarix #1
  * Time 2 months: Prevnar 13 #2, Hib #2
  * Time 3-4 months: Pediarix #2
  * Time 4-6 months: Draw post vaccine titers
  * Time 6-12 months: Administer Hepatitis #3 to patients not immunized prior to treatment for cancer, or with negative Hepatitis B titers after two immunizations.
  Other Names: vaccine, Prevnar 13; vaccine, Menactra II; Measles, mumps, rubella, MMR; Live, attenuated varicella vaccine, Varivax; Quadrivalent HPV Recombinant Vaccine
  Arms: A
Biological: Immunization Schedule patients > or = to 7 years and <11 years of age — * Time 0 months: Hib #1, Prevnar 13 #1, Hepatitis B #1
  * Time 1 month: Td#1, IPV #1(inactivated polio virus vaccine), Hepatitis B #2
  * Time 2-3 months: Prevnar 13 #2, Hib #2
  * Time 3-6 months: Td #2, Draw post vaccine titers Time 6-12 months: Administer Hepatitis #3 to patients not immunized prior to treatment for cancer, or with negative Hepatitis B titers after two immunizations.
  Other Names: vaccine, Prevnar 13; vaccine, Menactra II; Measles, mumps, rubella, MMR; Live, attenuated varicella vaccine, Varivax; Quadrivalent HPV Recombinant Vaccine
  Arms: B
Biological: Immunization Schedule patients > or = to 11 years of age — * Time 0 month: Hib#1, Prevnar 13#1, Hepatitis B #1
  * Time 1 month: Tdap(BOOSTRIX), Hepatitis B #2
  * Time 2-3 months: Hib #2, Prevnar 13#2, Menactra
  * Time 3-6 months: IPV, Draw post vaccine titers
  * Time 6-12 months: Gardasil (dose #2 given 2 months after first dose, and dose #3 given 6 months after first dose)
  Arms: C

SUMMARY:
This study will look at your body's response to the new immunizations. We want to see how well they will protect you. Immunization is the same as vaccination. Our goal is to protect you as much as we can. We do not want you to have the measles, mumps, or whooping cough. We are doing the study because there is no standard way to re-immunize people after cancer treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be < or less 18 years of age at cancer diagnosis
* Patient must be 3 to 24months following completion of chemotherapy for malignant disease.

  1. For patients <12 months following completion of therapy, CR must be documented within 3 months of enrollment.
  2. For patients >12 months, CR must be documented at approximately 12 months and then only as clinically indicated

  i. For patients with leukemia: bone marrow aspirate defined as <5% blasts, absence of cytogenetic abnormality by FISH or karyotype (if applicable) and no evidence of CSF involvement (if applicable) ii. For patients with solid tumors remission will be determined by appropriate radiologic scans, and other tests, including bone marrow aspirate and biopsies demonstrating absence of extrinsic cells and absence of specific FISH or cytogenetic abnormality (if applicable), iii. For patients with lymphoma, remission will be determined by bone marrow aspirate and biopsy, radiologic scans and other tests. Bone marrow will show <5% blasts, absence of cytogenetic abnormality by FISH or karyotype (if applicable), and flow cytometry (if lymphoma specific marker present) and absence of CNS disease by spinal fluid (if applicable)
* Patient may be of either gender and of any ethnic background
* Patients or their guardians must be able to understand the nature and risk of the proposed study and be able to sign consent.

Exclusion Criteria:

* Karnofsky score <70%.
* Female patients who are pregnant or lactating.
* Patients who have received an autologous or allogeneic HCT.
* Active uncontrolled bacterial or fungal infection.
* Patients who have a history of previous allergic reaction to vaccinations currently recommended by the ACIP.
* Patients on any immunosuppressive drugs.
* HIV-1,2 sero-positive patients.
* Patients or guardians not signing informed consent.
* Patients with prior allergic reaction to any vaccine component or to latex.
* Patients who have received Rituximab.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2007-07-10 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
To prospectively determine the response rate and duration of protective titers following revaccination with routine childhood immunizations in pediatric survivors of childhood cancer. | conclusion of study

SECONDARY OUTCOMES:
To determine whether in vitro parameters of lymphoid reconstitution correlate with response and duration of response. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Kernan, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org